CLINICAL TRIAL: NCT05375318
Title: BIOhabitats: Biological Validation of Vascular Habitats Within Astrocytoma Grade 4 at Molecular, Cellular, and Histopathological Levels
Acronym: BIOhabitats
Status: Completed | Type: Observational
Sponsor: Juan M Garcia-Gomez (Other)
Collaborators: Hospital Clínico Universitario de Valencia (Other); Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor-Investigator, Juan M Garcia-Gomez, Main Researcher. Head of Biomedical Data Science Lab at UPV, Universitat Politècnica de València
Organization: Universitat Politècnica de València (Other)
Other Study IDs: BIOhabitats
Record Dates: First submitted 2022-02-01; First posted 2022-05-16 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Astrocytoma, Grade IV; Glioblastoma; Glioblastoma Multiforme; Glioblastoma, IDH-wildtype; Glioblastoma, IDH-mutant; Glioblastoma IDH (Isocitrate Dehydrogenase) Wildtype; Glioblastoma IDH (Isocitrate Dehydrogenase) Mutant; High Grade Glioma
Keywords: Astrocytoma, Grade IV; vascularity; vascular habitats; ROIs; regions of interest; glioma segmentation; biological validation
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults patients with astrocytoma grade 4

SUMMARY:
The main purposes of this study are:

I. To assess that the four habitats within the tumor (HAT and LAT) and edema (IPE and VPE) in high-grade glioma are different at vascular, tissular, cellular and molecular levels.

II. To analyze the associations between the perfusion imaging markers and relevant molecular markers at the HTS habitats for high-grade glioma diagnosis, prognosis/aggressiveness, progression and/or prediction.

III. To analyze the associations between the perfusion imaging markers and immune markers at the HTS habitats useful in immunotherapy evaluation and/or patient selection.

IV. To prospectively validate the prognostic capacity (association with OS and PFS) and stratification capacity of the perfusion imaging markers calculated at the HTS habitats.

DETAILED DESCRIPTION:
High-grade glioma (HGG) are the most aggressive malignant primary brain tumor in adults with a median survival rate of 12-15 months. It still carries a poor prognosis despite aggressive treatment, which includes tumor resection followed by chemo-radiotherapy cycles. The inter-patient and intra-patient tumor heterogeneity is one of the responsible factors for the high aggressiveness of solid malignant tumors and their resistance against effective therapies.

Due to the extremely complex and heterogeneous biology of this tumor, the same treatment for all approach does not work well in this disease, and standard of care is not always the best option, calling for precision medicine to select the best therapeutic option in the right moment to each patient. This requires quantitative medical imaging, patient profiling, prognosis estimation, and expected response to treatment for objective decision making along with the patient management.

The Hemodynamic Tissue Signature (HTS) methodology, included in the ONCOhabitats site (www.oncohabitats.upv.es), provides an automated unsupervised method to describe the heterogeneity of the enhancing tumor and edema areas in terms of the angiogenic process located at these regions. HTS considers 4 habitats within the tumour: 1) the HAT habitat, which refers to the high angiogenic enhancing tumor part of the tumour, 2) the LAT habitat, which refers to the less angiogenic enhancing tumor area of the tumour, 2) the IPE habitat, which refers to the potentially infiltrated peripheral edema, and 4) the VPE habitat, which refers to the vasogenic peripheral edema of the tumour (Juan-Albarracin et al, 2016). Perfusion imaging markers, such as relative cerebral blood volume, can be calculated from these different vascular habitats, and they have been proven as clinically relevant for prognosis. The HTS methodology, as well as the prognostic capacity of these perfusion imaging markers, have been validated with a retrospective multicenter study that included 184 high-grade glioma patients from 7 European centers.

Furthermore, relevant associations have been found between the perfusion markers and clinical-routine biomarkers, such as IDH mutation, MGMT methylation (Fuster-Garcia et al, 2020), molecular subtype or microvessel area.

Considering these promising results and, in order to develop a decision support system based on pixel level Artificial Intelligent models for deciding treatment in high-grade glioma, it is necessary to develop a prospective study and to validate at biological level the vascular habitats defined by the HTS methodology.

The proposed objectives are based on the following hypothesis:

I. Since the tumor and edema HTS habitats (HAT, LAT, IPE and VPE) have been proven as different in relation to their hemodynamic and vascular behavior, the main hypothesis are that these are habitats are also significantly different at the vascular, tissular, cellular and molecular level.

II. Significant associations between the perfusion imaging markers calculated with the HTS methodology and both molecular and histopathological markers (useful in prognosis, monitoring and evaluation of therapies) have been found in previous studies. Therefore, the hypothesis are that relevant associations between the imaging markers and clinical-routine biomarkers, such as molecular and histopathological markers, exist.

III. Preliminary studies have shown associations between the perfusion imaging markers and molecular markers related with the immune action/suppression. In addition, previous works have demonstrated that immune and genomic correlates of response to immunotherapy treatments, such as anti-PD-1, in glioblastoma. Therefore, to find correlations between these immune and genomic signatures with perfusion imaging markers can be useful for decision making and evaluation of immunotherapies.

IV. Preliminary retrospective studies have demonstrated robust association between the perfusion imaging markers calculated at high and low angiogenic habitats and patient overall survival. These robust associations between the perfusion imaging markers and survival times will be demonstrated with a prospective study.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with Astrocitoma, Grade 4, cIMPACT-NOW: update 6 classification with histopathological/genetic confirmation who undergo the Stupp treatment

* Age > 18 years at diagnosis
* Patients with access to complete pre-operative MRI studies, including:

  * Pre gadolinium T1-weighted MRI
  * Post gadolinium T1-wighted MRI
  * T2-weighted MRI
  * T2-Fluid-Attenuated Inversion Recovery (FLAIR)
  * Dynamic Susceptibility Contrast (DSC) T2*-weighted perfusion sequences
  * Diffusion Weighted Imaging (DWI)
* Patients who undergo surgery with the possibility to collect samples from different regions of the tumor

Exclusion Criteria:

6

* Patient with congestive heart failure within 6 months prior to study entry (New York Heart Association >= Grade 3)
* Uncontrolled or significant cardiovascular disease, including:

  * Myocardial infarction and transient ischemic attack or stroke within 6 months prior to enrollment
  * Uncontrolled angina within 6 months
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  * Clinically significant abnormality on electrocardiogram (ECG)
* Pulmonary disease including or greater than grade 2 dyspnea or laryngeal edema, grade 3 pulmonary edema or pulmonary hypertension according to CTCAE 4.03

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with astrocytoma grade 4
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Molecular profile of each vascular habitat biopsied for each included patient | through study completion, an average of 1 year
  Molecular profile of each vascular habitat biopsied for each included patient, including main molecular alterations typically found in astrocytoma grade 4
Description at cellular level of each vascular habitat biopsied for each included patient, including cell types and cell density | through study completion, an average of 1 year
  Description at cellular level of each vascular habitat biopsied for each included patient, including cell types and cell density
Description at histopathological level of each vascular habitat biopsied for each included patient, including tissues, necrosis, vascularuture | through study completion, an average of 1 year
  Description at histopathological level of each vascular habitat biopsied for each included patient, including tissues, necrosis, vascularuture

CONTACTS AND LOCATIONS:
Locations (1):
- Biomedical Data Science Lab. Universitat Politècnica de València, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No